CLINICAL TRIAL: NCT02218489
Title: A Phase II, Double-Masked, Randomized, Vehicle-Controlled Study to Evaluate the Effect of KPI-121 0.25% Ophthalmic Suspension on Signs and Symptoms of Inflammatory Meibomian Gland Disease
Brief Title: Safety and Efficacy of KPI-121 in Subjects With Inflammatory Meibomian Gland Disease
Acronym: Maui
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-003
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Blepharitis
Keywords: Pain; Corticosteroid; Meibomian Gland Disease; Blepharitis; Eyelid; Ocular Discomfort
MeSH Terms: conditions — Blepharitis; Pain; Meibomian Gland Dysfunction | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle (placebo) dosed QID for up to 30 days in subjects with inflammatory meibomian gland disease
  Interventions: Drug: Vehicle
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator): KPI-121 0.25% Ophthalmic Suspension dosed QID for up to 30 days in subjects with inflammatory meibomian gland disease
  Interventions: Drug: KPI-121

INTERVENTIONS:
Drug: KPI-121 — KPI-121 drug product will be supplied in 0.25% strength as a suspension in opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate. Subjects randomized to placebo control arm will receive the same bottles containing all components at the concentrations used in the KPI-121 drug product with the exception of the active component, loteprednol etabonate.
  Other Names: KPI-121 0.25% Ophthalmic Suspension; Loteprednol etabonate
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: Vehicle — The vehicle control has the same composition as KPI-121 0.25% ophthalmic suspension except it does not contain loteprednol etabonate. The vehicle is essentially isotonic and is buffered to maintain pH 5.0 - 7.0. It is a sterile, aqueous solution supplied in the same white, low-density polyethylene plastic dropper bottle with the same white, controlled-drop polyethylene tip and white polypropylene closure as KPI-121 0.25% ophthalmic suspension.
  Other Names: KPI-121 0.25% Vehicle; Placebo
  Arms: Vehicle

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 ophthalmic suspension compared to vehicle (placebo) in subjects with signs and symptoms of inflammatory meibomian gland disease.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the efficacy and safety of KPI-121 ophthalmic suspension versus vehicle in subjects with signs and symptoms of inflammatory meibomian gland disease. The product will be studied over 28 days, with 1-2 drops instilled in each eye four times daily (QID).

ELIGIBILITY:
Inclusion Criteria:

Have a documented clinical diagnosis of inflammatory meibomian gland disease in both eyes.

Exclusion Criteria:

* Known hypersensitivity/contraindication to study product(s) or components.
* Be currently receiving treatment for glaucoma, have history of or current glaucoma, or an IOP (intraocular pressure) over 21mmHg at Visit 1 (Screening) or Visit 2 (Randomization).
* Be unwilling to discontinue warm compress therapy, lid expression, or lid massage 14 days prior to Day 1 and for the duration of the study.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; severe/serious systemic disease or uncontrolled medical condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within the 30 days prior to screening.
* Have had ocular surgery in the past 90 days or require ocular surgery during the study.
* In the opinion of Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Abrams, MD, Principal Investigator — Abrams Eye Center; Damien Goldberg, MD, Principal Investigator — Wolstan & Goldberg Eye Associates; Jodi Luchs, MD, Principal Investigator — South Shore Eye Center, LLP; Kelly Nichols, OD, PhD, Principal Investigator — UAB School of Optometry; Steven Rauchman, MD, Principal Investigator — North Valley Eye Medical Group; Kenneth Sall, MD, Principal Investigator — Sall Research Medical Center; John Sheppard, MD, Principal Investigator — Virginia Eye Consultants; Joseph Tauber, MD, Principal Investigator — Tauber Eye Center
Locations (8):
- United States (8):
  - UAB School of Optometry, Birmingham, Alabama
  - Sall Research Medical Center, Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Tauber Eye Center, Kansas City, Missouri
  - South Shore Eye Center, LLP, Wantagh, New York
  - Abrams Eye Center, Cleveland, Ohio
  - Virginia Eye Consultants, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 206 subjects were randomized, 1 of which were not included in any analysis population as the individual did not receive randomized treatment.
Groups:
- KPI-121 0.25% Ophthalmic Suspension: KPI-121 0.25% Ophthalmic Suspension dosed QID for up to 30 days in subjects with inflammatory meibomian gland disease
  KPI-121: KPI-121 drug product will be supplied in 0.25% strength as a suspension in opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
Period: Overall Study
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Started | 101 | 104
Completed | 96 | 101
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension | Total
Number analyzed (Participants) | 101 | 104 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (13.13) | 60.2 (11.28) | 59.4 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 134
  Male | 29 | 42 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 35 | 63
  Not Hispanic or Latino | 73 | 69 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 80 | 84 | 164
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 101 | 104 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Discomfort
Description: Comparison of change from baseline in ocular discomfort between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse at Visit 4 (Day 15).
Time Frame: Visit 2 (Day 1) to Visit 4 (Day 15)
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 101 | 104
score on a scale | -4.1 (13.8) | -2.4 (16.7)

2. Primary Outcome: Change From Baseline in Posterior Lid Margin Hyperemia in the Subgroup of Subjects With Greater Hyperemia at Baseline
Description: Comparison of change from baseline in posterior lid margin hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group in subjects with greater baseline hyperemia at Visit 4 (Day 15). The scale for posterior lid margin hyperemia was scored on a range from 0-4 with the following description:
  0=normal
  1. mild
  2. moderate
  3. severe
  4. very severe
Time Frame: Visit 2 (Day 1) to Visit 4 (Day 15)
Population: m1ITT- a subset of the ITT population with greater baseline hyperemia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 77 | 79
score on a scale | -0.5 (0.7) | -04 (0.7)

3. Secondary Outcome: Change From Baseline in Ocular Discomfort
Description: Comparison of change from baseline in ocular discomfort between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse at Visit 6 (Day 29).
Time Frame: Visit 2 (Day 1) to Visit 6 (Day 29)
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 101 | 104
score on a scale | -8.2 (17.1) | -5.0 (15.8)

4. Secondary Outcome: Change From Baseline in Posterior Lid Margin Hyperemia in the Subgroup of Subjects With Greater Hyperemia at Baseline
Description: Comparison of change from baseline in posterior lid margin hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group in the subgroup of subjects with greater hyperemia at baseline at Visit 6 (Day 29). The scale for posterior lid margin hyperemia was scored on a range from 0-4 with the following description:
  0=normal
  1. mild
  2. moderate
  3. severe
  4. very severe
Time Frame: Visit 2 (Day 1) to Visit 6 (Day 29)
Population: m1ITT- a subset of the ITT population with greater baseline hyperemia. m1ITT population minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 76 | 79
score on a scale | -0.4 (0.7) | -0.6 (0.7)

5. Secondary Outcome: Change From Baseline in Posterior Lid Margin Hyperemia
Description: Comparison of change from baseline in posterior lid margin hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group at Visit 4 (Day 15). The scale for posterior lid margin hyperemia was scored on a range from 0-4 with the following description:
  0=normal
  1. mild
  2. moderate
  3. severe
  4. very severe
Time Frame: Visit 2 (Day 1) to Visit 4 (Day 15)
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 101 | 104
score on a scale | -0.56 (0.72) | -0.55 (0.64)

6. Secondary Outcome: Change From Baseline in Posterior Lid Margin Hyperemia
Description: Comparison of change from baseline in posterior lid margin hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group at Visit 6 (Day 29). The scale for posterior lid margin hyperemia was scored on a range from 0-4 with the following description:
  0=normal
  1. mild
  2. moderate
  3. severe
  4. very severe
Time Frame: Visit 2 (Day 1) to Visit 6 (Day 29)
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 101 | 104
score on a scale | -0.63 (0.76) | -0.65 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a subject signed the informed consent at Visit 1 until they exited the study at Visit 6.
Arm/Group | Vehicle | KPI-121 0.25% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/104
Other Adverse Events (participants affected / at risk) | 8/101 | 8/104
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=101) | KPI-121 0.25% Ophthalmic Suspension (N=104)
Instillation site pain (General disorders) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor restricts the PI's rights to discuss or publish trial results until after the first to occur of the following:

(a) publication of such multi-center clinical trial results; (b) notification by sponsor that such a multi-center clinical trial submission is no longer planned; or ( c) the eighteen ( 18) month anniversary of the completion, abandonment or termination of such multi-center clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT02218489/Prot_SAP_000.pdf